CLINICAL TRIAL: NCT06062563
Title: An Exploratory Study to Evaluate the Efficacy of Anlotinib Hydrochloride Combined With Penpulimab in the Treatment of Radioiodine Refractory Differentiated Thyroid Cancer With First-line Resistance to Angiogenesis Inhibitors
Brief Title: Study of Anlotinib in Patients With Radioiodine Refractory Differentiated Thyroid Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T004
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced or Metastatic Radioiodine-refractory Differentiated Thyroid Carcinoma
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+ penpulimab (Experimental): Anlotinib：12 mg once daily for 2 weeks, followed by a rest of 1 week (21-day cycle)； Penpulimab：200mg Q3 W
  Interventions: Drug: Anlotinib Hydrochloride Capsule and Penpulimab

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule and Penpulimab — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor that inhibits both tumor angiogenesis and tumor cell proliferation by blocking VEGFR, FGFR, PDGFR, and c-Kit simultaneously.
  Penpulimab is a novel structure Immune checkpoint inhibitor. The combination of Penpulimab and RAI might have synergistic effects for DTC.
  Other Names: Anlotinib Hydrochloride Capsule; Penpulimab

SUMMARY:
This study aims to observe and explore the efficacy and safety of Anlotinib combined with penpulimab in the treatment of radioiodine refractory differentiated thyroid cancer with first-line resistance to angiogenesis inhibitors, and to summarize the treatment experience of population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined the study, signed the informed consent;
2. Patients were pathologically confirmed as locally advanced or metastatic differentiated thyroid cancer (DTC), having at least one measurable lesion (Response Evaluation Criteria In Solid Tumors (RECIST) 1.1);
3. Patients≥18 years of age; Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score: 0-2; Expected survival of more than 6 months;
4. Possessing imaging or clinical evidence of disease progression within the first 18 months of enrollment;
5. Progression of at least one anti-vascular drug（no more than 2）；
6. Tg and structural imaging examinations were performed at least twice before enrollment；
7. Meet any of the following while meeting the above 3 items:（1）Lesions were not iodine-avid；（2） The cumulative dose of RAI was ≥ 600 mCi or 22 GBq, with an interval of at least 3 months. （3） Radiographically documented disease progression within 18 months of RAI therapy despite the presence of iodine-131 affinity at the time of RAI therapy;
8. Major organ functions meet the following criteria within 7 days prior to the treatment:

   1. Hemoglobin (Hb) ≥90g/L;
   2. Absolute Neutrophil Count (ANC) ≥1.5×109/L;
   3. Platelet (PLT) ≥80×109/L；
   4. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);
   5. Alanine transferase (ALT) and Aspartate transferase (AST) ≤2.5×ULN; If accompanied by liver metastasis, ALT and AST ≤5×ULN； (f)Serum creatinine (Cr) ≤1.5×ULN or Creatinine clearance rate (CCr) ≥60ml/min； (g) The left ventricular ejection fraction was at least 50% of the normal level.
9. Female patients of reproductive age should agree that birth control (such as intrauterine device, birth control pills, or condoms) must be used during the study period and for six months after completion; Having a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating; Male patients should agree to use contraception during the study period and for six months after the end of the study.

Exclusion Criteria:

1. Complicated diseases and history:

   1. Histologic subtypes of thyroid cancer other than the differentiated type (e.g., medullary carcinoma, lymphoma, or sarcoma) could not be enrolled; Patients currently have or had other malignancies within 5years. Cured localized tumors could be enrolled（e.g., Skin basal cell carcinoma）
   2. Subjects with any severe and/or uncontrolled heart disease, including:

      1. According to the criteria of New York Heart Association (NYHA) grade II or above cardiac insufficiency or echocardiography: LVEF (left ventricular ejection fraction) <50%;
      2. Unstable angina
      3. A myocardial infarction had occurred within 1 year before the beginning of the treatment
      4. Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention
      5. QTc ≥450ms (male), QTc ≥470ms (female) (classified by New York heart association, NYHA);
2. Other anti-tumor treatment (including but not limited to chemotherapy, radiotherapy, etc.). were received within 28 days before the beginning of the treatment; TSH suppression therapy was excluded;
3. Patients who have previously used immune checkpoint inhibitors (including but not limited to nivolumab, pembrolizumab, toripalimab, sintilimab, etc.);

5) Patients with hypertension that was not falling to the normal range with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) were allowed to use antihypertensive treatment to achieve these parameters. Hypertensive crisis or hypertensive encephalopathy.

6) Multiple factors affect the absorption of oral drugs. 7）Patients at risk for gastrointestinal bleeding were not eligible, including the following: (1) patients with active peptic ulcer lesions and fecal occult blood (++); (2) patients with a history of melena and hematemesis within 3 months; 8). Active or uncontrolled severe infection (≥ Common Terminology Criteria for Adverse Events (CTC AE) 2 grade of infection); 9) Patients with concomitant diseases that, in the investigator's judgment, may seriously endanger patients' safety or may interfere with the completion of the study, or are deemed unsuitable for inclusion for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-11 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 2 years.
  The proportion of subjects who achieves a best overall response of CR(Complete Response) or PR(Partial response).
changes in Tg level | Baseline up to 2 years.
  The percentage of decrease in serum Tg from baseline;

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Baseline up to 2 years.
  From the first dose of Anlotinib to the date of objective disease progression or death, whichever occurs first
Disease-control Rate（DCR） | Baseline up to 2 years.
  The proportion of subjects response of CR, PR, or SD(Stable disease) (subjects achieving SD will be included in the DCR if they maintain SD for ≥4 weeks).
Duration of Response（DOR） | Baseline up to 2 years.
  From the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first.
Overall Survival（OS） | Baseline up to 2 years.
  From randomization to the time of death from any cause.
Time to response(TTR) | Baseline up to 2 years.
  From randomization to the time of response from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- YansongLin, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided